CLINICAL TRIAL: NCT05802550
Title: Metabo-lipidomic Analysis of the Ocular Surface and Aqueous Humor for the Search of Predictive Biomarkers of Ocular Surface Disease After Cataract Surgery: a Prospective Cohort Study
Brief Title: Metabo-lipidomics of the Ocular Surface for Cataract Surgery
Acronym: CATARACTOMIQUE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DR220231
Record Dates: First submitted 2023-03-13; First posted 2023-04-06 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Age-related Cataract
Keywords: Ocular surface; Cataract; Conjunctival impression cytology; Aqueous humor; Metabolomic; Lipidomic
MeSH Terms: conditions — Cataract | interventions — Interferometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Longitudinal cohort study in cataract patients (Other): Longitudinal, open-label, single-center cohort study in cataract patients.
  Interventions: Other: Ocular Surface Disease Index; Other: Interferometry; Other: Oxford score; Other: Conjunctival collection; Other: Aqueous humor collection; Other: Quantification of Tyndall and flare

INTERVENTIONS:
Other: Ocular Surface Disease Index — Questionnaire on ocular surface disorders
Other: Interferometry — Non-contact examination measuring NIBUT (non-invasive break-up time), meibography and tear meniscus measurement
Other: Oxford score — Investigation and quantification of superficial corneal punctate keratitis using the Oxford score
Other: Conjunctival collection — Two conjunctival prints: one for metabolomic and one for lipidomic
Other: Aqueous humor collection — Collection of 0.1 mL of aqueous humor immediately after making the accessory corneal incision at the beginning of the cataract surgery.
Other: Quantification of Tyndall and flare — Quantification of Tyndall and flare (from 1 to 4 crosses) in anterior chamber

SUMMARY:
Cataract is the world's leading cause of blindness, the treatment of which, exclusively surgical, offers excellent results in terms of visual recovery. It represents the most frequently performed surgery in France with more than 800,000 procedures each year. However, some patients develop postoperative ocular surface disease that can affect final visual acuity and quality of life. For example, dry eye disease, very common in the elderly, can be worsened by cataract surgery.

The identification of ocular surface biomarkers predictive of the postoperative risk of ocular surface disease carries the promise of better personalized perioperative care.

Conjunctival impression cytology represents a rapid, minimally invasive method of collecting conjunctival cells, which has proven its usefulness in the evaluation of diseases of the ocular surface. The aqueous humor is directly accessible at the beginning of the surgery.

An approach combining ultra-high performance liquid chromatography coupled with high-resolution mass spectrometry on the cells of the ocular surface and on the aqueous humor could improve our understanding of the physiopathology of ocular surface disease following cataract surgery.

This study will aim to 1) search for prognostic biomarkers of ocular surface disease after cataract surgery using a metabo-lipidomic approach 2) improve our understanding of the pathophysiological mechanisms involved.

ELIGIBILITY:
Inclusion criteria:

* Patient with cortico-nuclear and/or subcapsular cataract
* Age > or = 50 years
* Patient affiliated to a social security system
* Patient agreeing to participate in the study who provided his/her free and informed written consent

Exclusion criteria:

* History of ocular surgery or trauma (≤ 3 months)
* Other types of cataract excepted age-related or diabetic cataract
* Any eye drops or treatments that may interfere with the ocular surface
* Lens wearer
* Any general pathology with a known impact on the ocular surface (auto-immune disease, allergy)
* Proven allergy to povidone-iodine or to a component of the postoperative treatment
* Patient under legal protection (safeguard of justice, curatorship and guardianship), or in a situation of deprivation of freedom
* Patient unable to understand the nature and objectives of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative ocular surface disease | 1 months after cataract surgery
  Metabo-lipidomic analysis of intracellular content of the ocular surface preoperatively and aqueous humor intraoperatively to predict occurrence of ocular surface disease 1 month following cataract surgery.
Postoperative ocular surface disease | 3 months after cataract surgery
  Metabo-lipidomic analysis of intracellular content of the ocular surface preoperatively and aqueous humor intraoperatively to predict occurrence of ocular surface disease 3 months following cataract surgery.

SECONDARY OUTCOMES:
Change in number and semi-quantitative concentrations of ocular surface metabolites | From baseline to 1 month after cataract surgery
  Comparison of ocular surface metabolome using conjunctival impression cytology pre and postoperatively 1 month after cataract surgery
Change in number and semi-quantitative concentrations of ocular surface lipids | From baseline to 1 month after cataract surgery
  Comparison of ocular surface lipidome using conjunctival impression cytology pre and postoperatively 1 month after cataract surgery

CONTACTS AND LOCATIONS:
Locations (1):
- KHANNA, Tours, France

IPD SHARING:
Plan to Share IPD: No